CLINICAL TRIAL: NCT04646915
Title: Evaluation of Short-term Outcomes of Laparoscopic Radical Resection for Patients With Colon and Upper Rectum in Day Surgery Center
Brief Title: Evaluation of Short-term Outcomes of Day Surgery for Patients With CuRC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Clinical professor, West China Hospital
Other Study IDs: DS-CuRC-2020
Record Dates: First submitted 2020-11-11; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: day surgery; laparoscopic colectomy; laparoscopic anterior resection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CuRC undergoing day surgery: Patients with CuRC undergoing laparoscopic colectomy or anterior resection in day surgery center.
  Interventions: Other: Day surgery

INTERVENTIONS:
Other: Day surgery — Patients with CuRC who meet the standards will be assigned to day surgery center for surgery

SUMMARY:
To evaluate the feasibility and safety of laparoscopic colectomy and anterior resection for patients with colon/upper rectal cancer (CuRC) in day surgery center. Patients with colon or upper rectal cancer who meet the standards of day surgery will be enrolled, and laparoscopic radical resection of tumor will be performed in day surgery center. Perioperative outcomes of these patients and reasons for transferring to inpatient ward will be recorded prospectively.

DETAILED DESCRIPTION:
At present, with the development of laparoscopic surgery and the application of rapid rehabilitation, colorectal surgery has made great progress . At the same time, the application of evidence-based surgery and multimodal anesthesia in postoperative rehabilitation has accelerated the postoperative recovery. Moreover, several previous studies have shown that the implementation of ambulatory colorectal surgery can reduce the incidence of postoperative complications and shorten hospital stay. With the continuous development of rehabilitation surgery, the hospitalization time of colorectal surgery has been gradually shortened. In addition, studies had preliminarily proved the feasibility, safety and repeatability of outpatient colectomy and showed that 30% of patients with elective colectomy can be completed in outpatient department.

Therefore, the investigators designed the clinical pathway of day surgery for patients screened by outpatient department, so that these patients can complete laparoscopic radical resection of colon cancer or high rectal cancer in the day surgery center.

The aim of this study is to evaluate the feasibility and safety of day surgery center for patients with colon/upper rectal cancer (CuRC). Patients meet the inclusion criteria and exclusion criteria will be assigned to day surgery center to perform radically laparoscopic colectomy or anterior resection. Outcomes of interests including incidence of transfer to inpatient ward, readmission, perioperative adverse events will be recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients under 65 years old with colorectal cancer or patients older than 65 years assessed by anesthesiologist that their physical conditions were excellent;
2. Tumor located higher than 10cm by colonoscopy, and It is expected that the distal resection margin is above the peritoneal reflexes;
3. Tumor location was diagnosed clearly by abdominal CT, no severe local invasion required extensive resection, and no intraoperative colonoscopy was needed to determine the tumor site;
4. No distant metastasis assessed by preoperative imaging examination ；
5. There was no special abnormality in blood routine, blood biochemistry, blood coagulation, electrocardiogram and pulmonary function, and anesthesiologist assessed that the patient was safe for day surgery

Exclusion Criteria:

1. Patients with distant metastasis
2. Patients with ASA grade >Ⅲ and high risk in perioperative period are expected
3. Tumor was too small to clearly showed by abdominal CT, and Intraoperative colonoscopy is needed.
4. Patients who need neoadjuvant therapy (preoperative chemoradiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CuRC undergoning laparoscopic radical colectomy or anterior resection in day surgery center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of transfer to inpatient ward | one month after operation
  The incidence of patients who did not transfer to community hospital according to the plan after operation, and the causes of this situation.

SECONDARY OUTCOMES:
operation duration time | during the operation
  From the beginning of the skin incision to the end of the last incision was From the beginning of the skin incision to the end of the suture of last incision
Blood loss | during the operation
  intraoperative blood loss
Postoperative complications | 3 months after the surgery
  including incision infection，anastomotic leakage，respiratory infection, postoperative bleeding, and so on.
Length of Hospital stay (LOS) | 3 months after admission
  Time from admission to discharge
Costs of hospital expense | 3 months after admission
  Expense for disease treatment during hospitalization
Readmission rate | 90 days after surgery
  The proportion of patients who are re-hospitalized for postoperative adverse events within 90 days after discharge in all subjects.
Mortality | 90 days after surgery
  Death rate within 90 days after surgery in all patients after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, Study Chair — Department of Gastrointestinal Surgery, West China Hospital, Sichuan University
Locations (1):
- Guoxue Road 37#,West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided